CLINICAL TRIAL: NCT05975047
Title: A Phase 1a/1b Randomized, Double-Blind, Placebo-Controlled Study of Single and Multiple Ascending Doses of LIV001 in Healthy Subjects and Multiple Doses of LIV001 in Subjects with Mild-to-Moderate Active Ulcerative Colitis
Brief Title: A Study of LIV001 in Healthy Subjects and Those with Mild-to-Moderate Active Ulcerative Colitis (UC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Liveome Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: LIV001-01
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LIV001 (Experimental): Drug: LIV001
  Dosage level:
  Part A will receive single dose of either one or 10 capsules of 280 mg capsule of IP or placebo on Day 1; Part B participants will receive multiple doses of 280 mg capsule of IP or placebo from Day 1 to Day 14 after overnight fast ;
  Dosage form- capsule
  Route of administration- Oral
  Interventions: Drug: LIV001
- Placebo (Placebo Comparator): Placebo comparator taken by participants randomized to the placebo arm across Part A, B and C of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LIV001 — Part A- Participants will receive single dose of 280mg capsule on day 1 under fasting conditions; Part B- Participants will receive multiple doses of 280mg capsule from day 1 to day 14 under fasting conditions;
  Arms: LIV001
Drug: Placebo — Participants will receive matching placebo across Part A and B of the study
  Arms: Placebo

SUMMARY:
This study is only for the first in human phase 1a study designed to investigate the safety and tolerability of LIV001 in healthy participants. LIV001 will be investigated for the safety and efficacy in participants with Ulcerative Colitis (UC) in a phase 1b study.

DETAILED DESCRIPTION:
The study will be conducted in 2 parts. Approximately 36 subjects are planned to be enrolled into the study.

* In Part A (SAD), approximately 18 healthy subjects will be enrolled in 2 sequential cohorts (Cohorts SAD1 and SAD2) and randomized 2:1 to receive a single dose of investigational product (IP) (LIV001 or placebo)
* In Part B (MAD), approximately 18 healthy subjects will be enrolled into 2 sequential cohorts (Cohorts MAD1 and MAD2) and randomized 2:1 to receive LIV001 or placebo for 14 days.

Oversight of the study will be provided by a Safety review committee (SRC) comprising the Principal Investigator (PI), the local Medical Monitor (MM), and a representative of the Sponsor, at a minimum.

ELIGIBILITY:
Inclusion Criteria:

Part A (SAD) and Part B (MAD)

1. Male or female, aged 18 to 60 years (inclusive) at Screening.
2. Body mass index (BMI) 18 kg/m2 to ≤ 32 kg/m2 (inclusive) at Screening.
3. Subject is generally healthy, in the opinion of the Investigator, based on assessment of medical history, physical examination, vital signs, ECG, laboratory parameters, and other relevant tests conducted at Screening.
4. Subject has clinical laboratory values within normal range, as specified by the testing laboratory, at Screening and Day 1, unless deemed not clinically significant by the Investigator or delegate.
5. Nonsmoker or casual smoker who agrees to smoke ≤ 5 cigarettes per week (includes e-cigarettes and other nicotine and tobacco products) during the study, including follow-up, and is willing to abstain from smoking/nicotine products during the CTU confinement period(s) and for ≥ 5 days before each study visit.
6. Male and female must agree to contraceptive usage as per protocol from Screening through 90 days after final dose of IP.
7. Willing and able to comply with all study-related procedures and assessments, including attending visits to the CTU.
8. Able to read and understand, and willing to sign the ICF.
9. Willing to allow storage of blood and fecal samples for future studies of genetic make-up.

Exclusion Criteria:

Part A (SAD) and Part B (MAD)

1. Female subjects who are pregnant or lactating.
2. Abnormal ECG findings at Screening or Day -1 that are considered by the Investigator or designee to be clinically significant.
3. Has taken prescription medication (including antibiotics) within 14 days or over-the-counter (OTC) non-prescription medication, herbal remedies, vitamins or minerals, probiotics (foods containing probiotics are permitted), and yeast supplements (eg, Mutaflor®, Bioflor®) within 7 days prior to the first dose of IP that may, in the opinion of the Investigator, compromise subject safety or interfere with study procedures or data validity. Subjects may be rescreened after a washout period of 14 days for prescription medication or 7 days for OTC products. Use of oral contraceptives and paracetamol (1 to 2 therapeutic doses per week, ie, up to 2 g per week) and/or nonsteroidal anti-inflammatory drugs for symptomatic relief of minor symptoms is permitted.
4. Functional gastrointestinal disorders, eg, irritable bowel syndrome, functional heartburn, functional nausea, functional dyspepsia, functional constipation, and functional diarrhea.
5. Substance abuse-related disorder or a history of drug, alcohol (ie, regular use of > 21 units of alcohol per week) and/or substance abuse deemed significant by the Investigator.
6. Has taken any IP or received IP in another clinical trial within 30 days prior to the first dose of IP or 5 half-lives, whichever is longer.
7. History of significant hypersensitivity or severe allergic or anaphylactic reactions involving any drug (including ampicillin, clindamycin or imipenem), any constituent of the IP (LIV001 or its excipients), food or other precipitating agent (eg, bee sting). Subjects with clinically stable mild allergic conditions such as hay fever and mild eczema may be enrolled at the discretion of the Investigator.
8. Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus antibody (anti-HCV) at Screening.
9. Positive screen for drugs of abuse at Screening or Day -1, or positive screen for alcohol on Day -1.
10. Subject is, in the opinion of the Investigator, unlikely to comply with the clinical study protocol or is unsuitable for any other reason.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2023-09-24 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Upto 14 days from Part A; Upto 28 days for Part B
Number of participants with clinical laboratory abnormalities | Upto 14 days from Part A; Upto 28 days for Part B
Number of participants with changes in the 12-lead electrocardiogram (ECG) | Upto 14 days from Part A; Upto 28 days for Part B
Number of participants with changes in stools as self assessed through Bristol stool form scale (BSFS) | Upto 14 days from Part A; Upto 28 days for Part B

SECONDARY OUTCOMES:
Number of participants detected tection of LIV001 in stool samples by quantitative polymerase chain reaction (qPCR) | Upto 14 days from Part A; Upto 28 days for Part B

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Pty Ltd, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No